CLINICAL TRIAL: NCT03240289
Title: Use of Text Messaging to Reduce Barriers to Self-care for Low-income Pregnant Women With Diabetes
Brief Title: Texting for Diabetes Success in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00084353
Record Dates: First submitted 2017-07-14; First posted 2017-08-07 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Gestational Diabetes; Pregnancy in Diabetics
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy in Diabetics

STUDY DESIGN:
Intervention Model Description: Single arm feasibility and pilot testing study of a curriculum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Texting (Other): Texting group
  Interventions: Behavioral: Texting group

INTERVENTIONS:
Behavioral: Texting group — Women receive text messages to aid in their diabetes self-care tasks during pregnancy; these included appointment reminders, motivational messages, and nutrition/exercise tips.

SUMMARY:
Diabetes during pregnancy can be a challenging circumstance requiring extensive patient learning and self-care. The purpose of this study is to develop and pilot test a patient-centered diabetes education and self-care tool using text messaging to provide supportive messaging and education to underserved women with a pregnancy complicated by diabetes.

DETAILED DESCRIPTION:
Low-income, pregnant women in the Chicago area are frequently affected by obesity or diabetes. The addition of a disease in pregnancy amplifies the requirements for optimal self-care during pregnancy. This load of information poses a significant burden, particularly for women with additional socioeconomic barriers to self-care. Preliminary work suggests patients must overcome a number of social, psychological, and knowledge-based barriers to achieve successful diabetic control in pregnancy.

This project involves development and preliminary evaluation of a patient-centered education and self-care tool for use with women whose pregnancies are complicated by diabetes. The study begins with development of a text messaging curriculum to provide motivational and educational support. We will use a one-way, non-interactive text-based educational platform to provide supportive and educational messages to a cohort of 40 women with diabetes. Women receive 3-5 text messages per week until delivery. The goal is to develop a program that can be expanded to a clinical trial in which perinatal outcomes are assessed.

The primary outcome is patient satisfaction and opinions about the texting program, as measured via a qualitative interview upon study completion. Participants underwent an enrollment survey to assess health literacy/numeracy, diabetes self-efficacy, diabetes knowledge, personality, and social hassles. They underwent a baseline in-depth one-on-one interview focusing on barriers to successful self-care with pregnancy and diabetes. Follow-up surveys and an exit interview elicited information about their opinions of the texting program. Additional goals included determining feasibility for future expansion as a trial.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* English-speaking
* Have gestational diabetes mellitus, type 2 diabetes mellitus, or type 1 diabetes mellitus
* Age 18 years or older
* Access to a phone that can receive text messages

Exclusion Criteria:

* Gestational age greater than 30 weeks
* Women not meeting the above inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction and feedback | Up to 42 weeks
  A single qualitative interview of patient perspectives and areas for improvement in the text messaging program. Interview takes place between 35 weeks gestation and discharge after delivery (postpartum day 2)

SECONDARY OUTCOMES:
Diabetes self-efficacy (Measured using the Diabetes Empowerment Scale-Short Form) | Up to 42 weeks
  Assessment of diabetes self-efficacy. Survey takes place after 35 weeks gestation and before discharge after delivery (postpartum day 2)
Barriers and facilitators of diabetes self-management | Study enrollment
  Qualitative interview of patient experiences regarding having diabetes during pregnancy
Study feasibility (as measured by number of participants retained in the study) | Up to 42 weeks
  Ability to recruit and retain participants
Diabetes self-efficacy (Measured using the Perceived Diabetes Self-Management Scale) | Up to 42 weeks
  Assessment of diabetes self-efficacy. Survey takes place after 35 weeks gestation and before discharge after delivery (postpartum day 2)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Simon, MD, MPH, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: Undecided